CLINICAL TRIAL: NCT03300336
Title: Optimizing Function and Independence Through STRIDE (QUE 16-170)
Brief Title: Optimizing Function and Independence Through STRIDE
Acronym: STRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 16-015
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Early Ambulation
Keywords: Walking; Inpatients; Veterans; Early Ambulation; Quality of Life

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster Randomized Trial - a form of crossover design with unidirectional crossover (from control to experimental) but with randomization of when each cluster undertakes the transition. In the stepped wedge design, there is a staggered roll-out of the intervention, where the time and sequence of clusters that will start the intervention at each period determined by random allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Implementation of STRIDE program
  Interventions: Behavioral: STRIDE
- Usual Care (No Intervention): Pre-implementation before STRIDE program

INTERVENTIONS:
Behavioral: STRIDE — Implementation of STRIDE inpatient hospital mobility program
  Arms: Intervention

SUMMARY:
Optimizing Function and Independence Through STRIDE aims to implement the STRIDE inpatient hospital mobility program at 8 VAMC sites in a stepped-wedge design and evaluate patient outcomes before and after the program is implemented, as well as the efficacy of a usual vs enhanced implementation design.

DETAILED DESCRIPTION:
Background/Purpose. A key contributor to hospital-associated disability is immobility during hospitalization. While fewer than 5% of patients have physician orders for bed rest, hospitalized older adults spend only 3% of their time standing or walking. The hazards of immobility in the hospital have been recognized for more than two decades, but there are currently no VA-system wide approaches to address this important gap in clinical care.

STRIDE is a supervised inpatient walking program developed by an interdisciplinary team of investigators, clinicians and administrators at the Durham VA and funded by the VHA Office of GEC. STRIDE consists of a one-time gait and balance assessment conducted by a physical therapist, followed by daily supervised walks by a recreation therapy assistant for the duration of the hospital stay. Program evaluation has demonstrated high satisfaction among Veteran participants and reduced need for post-acute institutional care. As a result, the Durham VAMC funded STRIDE as a permanent program that currently serves over 650 Veterans annually, and the VHA Office of GEC funded a dissemination grant to launch the program at another medical center. The investigators' initial experience with STRIDE implementation suggests interprofessional relationships and team dynamics are key determinants to the success of a new hospital-based clinical program that requires collaborative processes involving multiple disciplines.

As part of the investigators' Optimizing Function and Independence QUERI, the investigators plan to implement the STRIDE clinical program at 8 VAMC sites in a stepped-wedge design with sites randomized to implementation strategy and start date.

Objectives. The investigators plan to conduct an evaluation to examine the impact of STRIDE on patient outcomes.

Key questions: Do STRIDE participants have fewer discharges to skilled nursing facilities and shorter lengths of stay? Do STRIDE participants have better physical function and higher health-related quality of life at 30 days post-discharge? What is the value of STRIDE from the Veteran's perspective? The investigators also plan to conduct a mixed method evaluation that examines implementation outcomes and provider team experience that will not be reported here.

Methodology. The investigators will compare patients discharged from sites before and after the STRIDE program is implemented to assess discharge to skilled nursing facilities and length of stay (approx. n=2000). A subset of patients participating in the STRIDE program and a comparison group will be surveyed 30 days post-hospital discharge to assess outcomes including health status, physical function, and quality of life. A subset of patients will be interviewed one week post-discharge to gain feedback about the STRIDE program and perceived benefits of a hospital inpatient mobility program.

In 2023, the following updates were made after results were initially uploaded to clinical trials as follows: primary outcome description and results were modified to reflect discharge to skilled nursing facility versus discharge to home and modifications were made to the sample and discharge to skilled nursing home and length of stay outcomes due to receipt of more complete data sources for use to determine eligibility and to assess the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

Inclusion/Exclusion listed here apply to subset of patients providing consent for telephone interviews:

* Able and willing to provide informed consent (does not lack decision-making capacity)
* Discharged from a participating hospital within the preceding 30 days
* Age >= 60
* Index admission for medical illness
* Community-dwelling (i.e. not in a nursing home or institutional care) prior to hospital visit
* Ability to ambulate safely and independently (does not need help walking across a small room)
* Valid telephone number in the medical record
* Admitted to a STRIDE ward and discharged from a STRIDE ward
* Index hospital stay was in a ward identified to participate in the STRIDE program

Exclusion Criteria:

* Patient deceased
* Index hospital stay was < 2 business days
* Currently hospitalized
* Current high-risk suicide flag in medical record
* Diagnosis of cognitive impairment or dementia
* Difficulty with or unable to communicate on the telephone, or no telephone access
* Discharged to another hospital or acute care setting
* Transferred into index hospital from another hospital
* Bedrest order not lifted for at least 2 days on STRIDE ward

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13857 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2021-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan N. Hastings, MD MHSc, Principal Investigator — Durham VA Medical Center, Durham, NC; Courtney H Van Houtven, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC; Virginia Wang, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be available upon request. Prior to distribution, a local privacy officer and study statistician will certify that the dataset contains no protected health information (PHI). Data will be provided to requestor in electronic format.
  Sufficient data and descriptors will be made available to duplicate statistical analysis and confirm conclusions in publication.
  No data or statistical code that could lead to re-identification of individuals will be released.
  Data will be stored & maintained in an approved, secured location as described in the VA Research Data Inventory Form.
  The study statistician will create de-identified, publication-specific datasets that includes all variables presented in the study publication.
  Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re-identify any individual whose data are included in the dataset.
Time Frame: Available upon request.
Access Criteria: Data will only be released per appropriate authorizations or agreements. Written agreements will specify that recipients are prohibited from taking steps to re- identify any individual whose data are included in the dataset.

REFERENCES:
- [Derived] Kaufman BG, Hastings SN, Meyer C, Stechuchak KM, Choate A, Decosimo K, Sullivan C, Wang V, Allen KD, Van Houtven CH. The business case for hospital mobility programs in the veterans health care system: Results from multi-hospital implementation of the STRIDE program. Health Serv Res. 2024 Dec;59 Suppl 2(Suppl 2):e14307. doi: 10.1111/1475-6773.14307. Epub 2024 Apr 17. PMID 38632179
- [Derived] Hastings SN, Stechuchak KM, Choate A, Van Houtven CH, Allen KD, Wang V, Colon-Emeric C, Jackson GL, Damush TM, Meyer C, Kappler CB, Hoenig H, Sperber N, Coffman CJ. Effects of Implementation of a Supervised Walking Program in Veterans Affairs Hospitals : A Stepped-Wedge, Cluster Randomized Trial. Ann Intern Med. 2023 Jun;176(6):743-750. doi: 10.7326/M22-3679. Epub 2023 Jun 6. PMID 37276590
- [Derived] Wang V, D'Adolf J, Decosimo K, Robinson K, Choate A, Bruening R, Sperber N, Mahanna E, Van Houtven CH, Allen KD, Colon-Emeric C, Damush TM, Hastings SN. Adapting to CONNECT: modifying a nursing home-based team-building intervention to improve hospital care team interactions, functioning, and implementation readiness. BMC Health Serv Res. 2022 Jul 29;22(1):968. doi: 10.1186/s12913-022-08270-1. PMID 35906589
- [Derived] Hastings SN, Stechuchak KM, Choate A, Mahanna EP, Van Houtven C, Allen KD, Wang V, Sperber N, Zullig L, Bosworth HB, Coffman CJ. Implementation of a stepped wedge cluster randomized trial to evaluate a hospital mobility program. Trials. 2020 Oct 16;21(1):863. doi: 10.1186/s13063-020-04764-7. PMID 33076997
- [Derived] Wang V, Allen K, Van Houtven CH, Coffman C, Sperber N, Mahanna EP, Colon-Emeric C, Hoenig H, Jackson GL, Damush TM, Price E, Hastings SN. Supporting teams to optimize function and independence in Veterans: a multi-study program and mixed methods protocol. Implement Sci. 2018 Apr 20;13(1):58. doi: 10.1186/s13012-018-0748-3. PMID 29678137
- See also: Function QUERI program — https://www.queri.research.va.gov/programs/function.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 7134 | 6723
Completed | 7134 | 6723
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patient-hospitalizations
Units Other Than Participants: patient hospitalizations
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 7134 | 6723 | 13857
Number analyzed (patient hospitalizations) | 9070 | 8167 | 17237
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.0 (8.6) | 72.8 (8.8) | 72.9 (8.7)
Sex: Female, Male [Count of Units; unit: patient hospitalizations]
  Female | 308 | 213 | 521
  Male | 8762 | 7954 | 16716
Ethnicity (NIH/OMB) [Count of Units; unit: patient hospitalizations]
  Hispanic or Latino | 157 | 435 | 592
  Not Hispanic or Latino | 8751 | 7626 | 16377
  Unknown or Not Reported | 162 | 106 | 268
Race (NIH/OMB) [Count of Units; unit: patient hospitalizations]
  American Indian or Alaska Native | 56 | 46 | 102
  Asian | 10 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 43 | 53 | 96
  Black or African American | 2468 | 2418 | 4886
  White | 6206 | 5417 | 11623
  More than one race | 70 | 91 | 161
  Unknown or Not Reported | 217 | 135 | 352
Region of Enrollment [Number; unit: patient hospitalizations]
  United States | 9070 | 8167 | 17237

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Discharged to Skilled Nursing Facility
Description: Discharge to skilled nursing facility (versus home) will be assessed via administrative data pulls and chart review (not patient report).
Time Frame: Assessed at hospital discharge, an average of 7 days
Population: Discharge to skilled nursing facility was analyzed for the first hospitalization for each patient during the study period. Patients can be in both intervention and usual care groups if hospitalized during the respective intervention and usual care time periods; however, for this outcome patients will be analyzed in only one group, based upon the earliest of their hospitalizations if had more than one.
Measure: Mean (Standard Error); unit: proportion of patients
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 6141 | 6722
proportion of patients | 0.16 (0.02) | 0.20 (0.03)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the 7 post-baseline timepoints), and a site-level random effect. Model was not adjusted for patient characteristics. Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.01, generalized linear model — a priori threshold for statistical significance p <.05; generalized linear model with a logit link and a binomial distribution; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.64 to 0.93] — Odds in intervention numerator vs odds in usual care denominator

2. Primary Outcome: Hospital Length of Stay (Days)
Description: Hospital length of stay will be assessed via administrative data pulls (not patient report)
Time Frame: Assessed at hospital discharge, an average of 7 days
Population: Length of stay was analyzed for the first hospitalization for each patient during the study period. Patients can be in both intervention and usual care groups if hospitalized during the respective intervention and usual care time periods; however, for this outcome patients will be analyzed in only one group, based upon the earliest of their hospitalizations if had more than one.
Measure: Mean (Standard Error); unit: Days
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 6141 | 6722
Days | 6.92 (0.21) | 6.58 (0.20)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the 7 post-baseline time points), a site-level random effect and random effects for each of the time periods. Model was not adjusted for patient characteristics. Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.25, generalized linear model — a priori threshold for statistical significance p<.05; generalized linear model with a log link and negative binomial distribution; rate ratio = 1.05, 95% CI 2-sided [0.97 to 1.15] — The rate ratio compares the intervention rate in the numerator vs the usual care rate in the denominator

3. Secondary Outcome: Patient Physical Function - Disability
Description: Analysis of physical function will be measured by the Late Life Function and Disability Instrument (LL-FDI) - Disability Component. Raw scores transformed to scaled scores ranging from 0-100, with higher scores reflecting higher functioning.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: Veterans completing a telephone survey 30 days after discharge from an eligible hospitalization. While Veterans may have multiple eligible hospitalizations, in the study framework Veterans can only be surveyed once.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 67.31 (1.55) | 65.99 (1.39)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care group: 5 out of 227 Missing data due to item nonresponse in intervention group: 18 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.52, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = 1.32, 95% CI 2-sided [-2.70 to 5.33] — Estimated difference calculated as intervention minus control

4. Secondary Outcome: Patient Physical Function - Limitations
Description: Analysis of physical function will be measured by the Late Life Function and Disability Instrument (LL-FDI) - Limitations Component -Instrumental Role Domain. Raw scores transformed to scaled scores ranging from 0-100, with higher scores reflecting higher functioning.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 65.67 (1.84) | 64.12 (1.66)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.66, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = 1.56, 95% CI 2-sided [-3.14 to 6.25] — Estimated difference calculated as intervention minus control

5. Secondary Outcome: Patient Physical Function
Description: Analysis of physical function will be measured by the Late Life Function and Disability Instrument (LL-FDI) - Function Component - Basic Lower Extremity Functioning Domain. Raw scores transformed to scaled scores ranging from 0-100, with higher scores reflecting higher functioning.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: Patient telephone survey 30 days post discharge
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 67.88 (1.64) | 68.40 (1.50)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect.. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care group: 5 out of 227 Missing data due to item nonresponse in intervention group: 14 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.81, Mixed Models Analysis — a priori threshold for significance p<.05; Mean Difference (Net) = -0.52, 95% CI 2-sided [-4.74 to 3.70] — Estimated difference calculated as intervention minus control

6. Secondary Outcome: Proportion Highly Satisfied With Care
Description: Analysis of satisfaction with care will be measured with the Consumer Assessment of Healthcare Providers and Systems (CAHPS)-based item "Would you recommend this hospital to other Veterans if they needed care for a condition such as yours?" Responses were categorized into two categories: highly satisfied (responses of "Definitely Yes") and less satisfied (responses of "Probably Yes", "Probably No", and "Definitely No").
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: proportion of patients
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
proportion of patients | 0.85 (0.04) | 0.84 (0.04)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 0 out of 227 Missing data due to item nonresponse in intervention: 5 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.74, generalized linear model — a priori threshold for statistical significance p<.05; generalized linear model with a logit link and a binomial distribution; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.55 to 2.32] — Odds in intervention numerator vs odds in usual care denominator

7. Secondary Outcome: Health Utility
Description: Analysis of health utility, a health-related quality of life measure, will be assessed with the ICEpop CAPability measure for adults (ICECAP-A). Tariff values for an overall state are calculated by summing the values across the individual attributes (Feeling settled and secure; Love, friendship and support; Being independent; Achievement and progress; and Enjoyment and pleasure). Tariff values can range from 0 to 1, with higher values reflecting greater quality of life.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: Patients completing a telephone survey 30 days post discharge
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 0.82 (0.02) | 0.80 (0.01)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 14 out of 227 Missing data due to item nonresponse in intervention: 33 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.40, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.03 to 0.06] — Estimated difference calculated as intervention minus control

8. Secondary Outcome: Health-related Quality of Life
Description: Analysis of health-related quality of life will be measured by the Euroqol (EQ-5D). Response profiles are mapped to a score via a crosswalk. Scores range from -0.109 to 1.0, with higher scores reflecting a higher quality of life.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 0.76 (0.02) | 0.73 (0.02)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 7 out of 227 Missing data due to item nonresponse in intervention: 23 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.18, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.01 to 0.07] — Estimated difference calculated as intervention minus control

9. Secondary Outcome: Mobility in the Environment
Description: Analysis of mobility in the environment will be assessed by the Life Space Questionnaire. The composite score incorporates use of equipment, need for personal help, and frequency of movement. Scores range from 0-120 with higher scores reflecting greater mobility.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 58.81 (3.26) | 58.01 (3.02)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 1 out of 227 Missing data due to item nonresponse in intervention: 4 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.83, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = 0.80, 95% CI 2-sided [-6.38 to 7.98] — Estimated difference calculated as intervention minus control

10. Other Pre Specified Outcome: Sleep
Description: Analysis of sleep functioning will be assessed with the sleep subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS-29). Raw scores converted to t-scores ranging from 32.0 to 73.3. Higher scores indicate more sleep disturbance.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 51.79 (0.98) | 50.33 (0.90)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 2 out of 227 Missing data due to item nonresponse in intervention: 6 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.25, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = 1.46, 95% CI 2-sided [-1.05 to 3.96] — Estimated difference calculated as intervention minus control

11. Other Pre Specified Outcome: Proportion of Participants Self-reporting at Least One Fall
Description: Veterans self-reporting at least one fall in the 30 days since discharge from an eligible hospitalization, as queried during a telephone survey.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: proportion of patients
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
proportion of patients | 0.18 (0.02) | 0.16 (0.03)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 1 out of 227 Missing data due to item nonresponse in intervention: 3 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.59, generalized linear model — a priori threshold for statistical significance p<.05; generalized linear model with a logit link and a binomial distribution; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.68 to 1.99] — Odds in intervention numerator vs odds in usual care denominator

12. Other Pre Specified Outcome: PROMIS-29 Pain Subscale
Description: Analysis of pain will be assessed with the pain subscale of the Patient-Reported Outcomes Measurement Information System (PROMIS-29). Raw scores converted to t-scores ranging from 41.6 to 75.6. Higher scores indicate higher (worse) pain interference.
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 56.46 (0.96) | 55.47 (0.91)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 11 out of 227 Missing data due to item nonresponse in intervention: 20 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.47, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = 0.99, 95% CI 2-sided [-1.71 to 3.69] — Estimated difference calculated as intervention minus control

13. Other Pre Specified Outcome: Depression
Description: Analysis of depression will be assessed with the Center for Epidemiologic Studies Depression Scale (CESD-10). Scores range from 0-30, with higher scores reflecting more depressive symptoms
Time Frame: 30 days following hospital discharge, hospital stay an average of 6 days
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 399 | 227
score on a scale | 9.04 (0.57) | 9.11 (0.53)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Model included a time-varying indicator for when STRIDE program launched, fixed effects for time (indicator variables for each of the time periods) and a site-level random effect. Model was not adjusted for patient characteristics. Missing data due to item nonresponse in usual care: 2 out of 227 Missing data due to item nonresponse in intervention group: 7 out of 399 Estimated means and standard errors are provided in Outcome Measure Data table; Test type: Superiority; p = 0.94, Mixed Models Analysis — a priori threshold for statistical significance p<.05; Mean Difference (Net) = -0.07, 95% CI 2-sided [-1.76 to 1.62] — Estimated difference calculated as intervention minus control

ADVERSE EVENTS:
Time Frame: 6 months post discharge, hospital stay an average of 7 days
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/7134 | 0/6723
Serious Adverse Events (participants affected / at risk) | 0/7134 | 0/6723
Other Adverse Events (participants affected / at risk) | 0/7134 | 0/6723

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT03300336/Prot_SAP_000.pdf